CLINICAL TRIAL: NCT03087253
Title: Prospective Multicenter Natural History Study of Lipodystrophy Syndromes to Determine Prevalence, Incidence and Predictors of Diabetes and Severe Hypertriglyceridemia, and Their Complications
Brief Title: The LD Lync Study - Natural History Study of Lipodystrophy Syndromes
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elif Oral, Professor of Medicine, University of Michigan
Other Study IDs: HUM00127427
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Lipodystrophy (Genetic or Acquired, Non HIV)
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Genetic lipodystrophy syndromes are extremely rare, orphan diseases with overall estimated prevalence of less than 2,000 in the United States. These rare disorders characterized by selective loss of adipose tissue and predisposition to insulin resistance and its metabolic complications diabetes, dyslipidemia and hepatic steatosis. Due to these metabolic problems, atherosclerotic vascular disease, recurrent episodes of acute pancreatitis, cirrhosis and other morbidities complicate the lives of these patients.

In the last few years, several genes for CGL (AGPAT2, BSCL2, CAV1 and PTRF); FPL (LMNA, PPARG, AKT2, CIDEC, LIPE, PLIN1, PCYT1A and ADRA2A); MAD (LMNA and ZMPSTE24); APS (LMNA); autoinflammatory (PSMB8); NPS (FBN1, CAV1); SHORT syndrome (PIK3R1); and MDP syndrome (POLD1) have been identified. However, there is paucity of information about the natural history of these rare syndromes, especially genotype-specific causes of morbidity and mortality.

To overcome the problems outlined above, this multicenter, collaborative, prospective, observational natural history cohort study will be conducted on approximately 500 patients with genetic or acquired lipodystrophy syndromes. Patients will be assessed on a yearly basis for approximately 5 to 7 years to collect robust clinical, metabolic, morbidity and mortality data. Medical history and patient questionnaires will be completed on a yearly basis by patients registered in the study. Clinical data such as vitals, laboratory results and anthropometric measurements will also be collected from patients' medical records if available.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of genetic lipodystrophy Supportive data: 1) Presence of biallelic known disease-causing variants in the genes for autosomal recessive lipodystrophy syndromes; 2) Presence of a known (or de novo loss of function) disease-causing variant in the genes for autosomal dominant lipodystrophy syndromes.

Exclusion Criteria:

* HIV-infected patients with lipodystrophy
* Drug-induced lipodystrophy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a clinical diagnosis of genetic lipodystrophy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of diabetes mellitus | 4 years
  Number of subjects with diabetes mellitus or who develop diabetes mellitus

SECONDARY OUTCOMES:
Prevalence of severe hypertriglyceridemia | 4 years
  Number of subjects with severe hypertriglyceridemia (greater than 500 md/dL) or who develop severe hypertriglyceridemia
Incidence of severe morbidities and causes of mortality | 4 years
  Incidence of severe morbidities (acute pancreatitis, congestive heart failure, cirrhosis, liver failure) and causes of mortality in subjects

CONTACTS AND LOCATIONS:
Overall Officials: Elif A Oral, MD, Principal Investigator — Professor of Medicine
Locations (3):
- United States (2):
  - National Institutes of Health, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided